CLINICAL TRIAL: NCT05745519
Title: Discussion on Pulse Diagnosis and Heart Rhythm Variability of Patients With Chronic Insomnia
Status: Completed | Type: Observational
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20220101
Record Dates: First submitted 2023-02-16; First posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Heart Rate Variability; Insomnia Chronic
Keywords: Insomnia; Pulse; Heart rate variability
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The experimental group: Aged 40-79 years old, complained of insomnia symptoms in the past month, at least three times a week, for a month, such as: difficulty falling asleep, waking up in the middle of the night, waking up unable to fall asleep, waking up in the morning and still not getting enough sleep
  Interventions: Other: Pittsburgh sleep quality index (PSQI); Device: ANSWatch
- The control group: Healthy volunteer subjects aged 40-79 without insomnia.
  Interventions: Other: Pittsburgh sleep quality index (PSQI); Device: ANSWatch

INTERVENTIONS:
Other: Pittsburgh sleep quality index (PSQI) — The scale is suitable for the evaluation of sleep quality in patients with sleep disorders and mental disorders, as well as for the evaluation of sleep quality in general people.
Device: ANSWatch — Measure eight physiological parameters including heartbeat, systolic blood pressure, diastolic blood pressure, heart rhythm variability HRV, low frequency component LF, high frequency component HF, LF/HF low frequency high frequency component ratio, and irregular heartbeat within five minutes

SUMMARY:
Discuss the objective assessment of patients with insomnia by pulse diagnosis, and measure by subjective questionnaire and physiological instruments.

DETAILED DESCRIPTION:
In Taiwan, insomnia is a prevalent illness. Clinical symptoms of sleep disturbances are rather typical now that the epidemic has taken hold. Pulse diagnosis is an important diagnostic method for insomnia in traditional Chinese medicine(TCM). TCM pulse diagnosis is not yet a widely used clinical diagnostic method for illnesses, nevertheless. Clinical use and teaching should benefit greatly if pulse diagnosis or learning can be made more objective or data-based.

ELIGIBILITY:
Inclusion Criteria:

* aged 40-60 years
* Complaints of insomnia symptoms in the past month that lasted for at least one week, such as difficulty falling asleep, waking up easily in the middle of the night, unable to fall asleep after waking up, still not getting enough sleep after waking up in the morning
* The score of sleep disorder on the Pittsburgh Sleep Quality Scale was more than 5 points

Exclusion Criteria:

* History of psychiatric disorders
* History of sleep apnea or nocturnal myoclonus
* Center or neurodegenerative disease
* Cancer
* Melatonin or sleeping pills use in the past month

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In the experimental group, select subjects who meet the following conditions: aged 40-79 years, who complained of insomnia symptoms in the past month, at least three times a week for one month, such as: difficulty falling asleep, waking up in the middle of the night, unable to wake up Falling asleep, waking up in the morning still feeling sleepy. Control group: healthy voluntary subjects aged 40-79 without insomnia.
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Pittsburgh sleep quality index (PSQI) | 15 minutes
  Pittsburgh sleep quality index (PSQI)

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | 15 minutes
  The Hospital Anxiety and Depression Scale (HADS) is a self-assessment questionnaire that has been found to be a reliable instrument for detecting states of anxiety and depression in the setting of hospital outpatient clinic.
Epworth Sleepiness Scale (ESS) | 15 minutes
  The ESS is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3), their usual chances of dozing off or falling asleep while engaged in eight different activities
The Green Climacteric Scale(GCS) | 15 minutes
  The Menopausal Symptom Scale will be used to measure menopausal symptoms in women. This scale was developed by Greene, with 21 items and four subscales: psychological, physiological, vasomotor, sexual dysfunction and other symptoms
General Sleep Disturbance Scale(GSDS) | 15 minutes
  Measure the patient's non-cognitive symptoms, family caregivers' perceived negative feelings of stress, caregivers' depression and sleep disturbance.
Constitution in Chinese Medicine Questionnaire (CCMQ) | 15 minutes
  The Chinese Medicine Constitutional Questionnaire (CCMQ) was developed by Wang et al. in Mainland China, according to the consensus of experts on types of BC TCM. It has 60 items measuring 9 types of BC:
  soft, lacking qi, lacking yang, lacking yin, moist sputum, moist heat, blood stasis, impaired qi and especially visceral organs. It was tested in the Beijing population to establish its facial validity. Its reliability and construction value have been proven in 2500 people from five different geographical districts in China

CONTACTS AND LOCATIONS:
Locations (1):
- Ministry of Health and Welfare Tainan Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided